CLINICAL TRIAL: NCT03479528
Title: The Predictive Value of Alarm Symptoms in Patients With Dyspepsia Based on Roman IV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Collaborators: Xijing Hospital (Other); Tang-Du Hospital (Other); Xi'an No.3 Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018013
Record Dates: First submitted 2018-03-08; First posted 2018-03-27 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-02

CONDITIONS: Dyspepsia
Keywords: Dyspepsia,alarm symptoms，Roman IV
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dyspepsia: All patients who were satisfied with the inclusion criteria and exclusion criteria in the department of the second affiliated hospital of Xi'an jiaotong university,Xijing Hospital, Tangdu Hospital, Xi'an No.3 Hospital, and received investigation.

SUMMARY:
Functional dyspepsia is one of the most common gastrointestinal disorders (FGIDs) encountered in clinical practice.Clinical diagnosis is notoriously unreliable in diagnosing the underlying cause of dyspepsia,but a number of alarm features have been suggested as indicating patients at higher risk for serious disease. The predictive value of alarm symptoms still require more researches. Rome IV introduced more precisely define the minimal thresholds for frequency and severity of each individual symptom, primarily for scientific purposes,but data still need to be collected to define thresholds based on the frequency and/or severity of symptoms that impair quality of life.A cross-sectional study was conducted to assess the predictive value of alarm symptoms in patients with dyspepsia based on Roman IV.Through endoscopy results to determine whether dyspepsia is organic or functional, benign or malignant, through contacts with the basic data, to determine the alarm symptoms

DETAILED DESCRIPTION:
Functional dyspepsia is one of the most common gastrointestinal disorders (FGIDs) encountered in clinical practice. Functional dyspepsia is a clinical syndrome characterized by chronic and recurrent gastroduodenal symptoms in the absence of any organic or metabolic disease that is likely to explain the symptoms.Functional dyspepsia has a high incidence in the population.Clinical diagnosis is notoriously unreliable in diagnosing the underlying cause of dyspepsia,but a number of alarm features have been suggested as indicating patients at higher risk for serious disease.However, previous studies noted that the sensitivity of alarm features for predicting cases with upper GI malignancies is unsatisfactory. The predictive value of alarm symptoms still require more researches. Rome IV was introduced in 2016. Rome IV introduced more precisely define the minimal thresholds for frequency and severity of each individual symptom, primarily for scientific purposes,but data still need to be collected to define thresholds based on the frequency and/or severity of symptoms that impair quality of life.A cross-sectional study was conducted to assess the predictive value of alarm symptoms in patients with dyspepsia based on Roman IV.All patients who were satisfied with the inclusion criteria and exclusion criteria in the department of the second affiliated hospital of Xi'an jiaotong university, Xijing Hospital, Tangdu Hospital, Xi'an No.3 Hospital, and received investigation.Inclusion criteria included:Symptoms of upper digestive tract for more than 6 months or 3 monthes（postprandial fullness, early satiation,epigastric pain, and epigastric burning）;Older than 18;From March 2018 to January 2011，received gastroscope and upper abdominal B ultrasound examination;agreeing the informed consent.Data collection:Basic information：name, age, height, weight, gender, marriage;Dyspepsia: symptoms of indigestion, duration of indigestion, and weekly incidence of indigestion;Abnormal symptoms: weight loss, anemia, anorexia, vomiting, blackstool, dysphagia;Lifestyle habits: spicy food, smoking, drinking, sleep quality, daily exercise time;Family history, helicobacter pylori infection, abdominal color ultrasound results,Cost.Through endoscopy results to determine whether dyspepsia is organic or functional, benign or malignant, through contacts with the basic data, to determine the alarm symptoms.Further more, this study was proved by the ethical committee of second hospital of Xi'an jiaotong university.

ELIGIBILITY:
Inclusion criteria:

1. Aged 18 years and older;
2. Presence of dyspeptic symptoms according with Rome IV criteria (Discomfort was characterized by the presence of one or more symptoms that included bothersome postprandial fullness, bothersome early satiation, bothersome epigastric pain, bothersome epigastric burning, Symptoms had to be present for at least 3 months within the preceding 6 months);
3. From March 2018 to January 2019, patient went to the Gastroenterology clinics of the second affiliated hospital of xi'an jiaotong university, Xijing Hospital, Tangdu Hospital, Xi'an No.3 Hospital, and received gastroscopy;
4. Upper abdominal ultrasonography, blood routine examination, liver function test were conducted within six months.

Exclusion criteria:

1. History of esophagitis or ulcer disease or other organic upper gastrointestinal disease, pancreaticobiliary disease, metabolic disease(abnormal thyroid function, diabetes );
2. Were pregnant, might become pregnant, or were lactating;
3. Major abdominal surgery;
4. Severe neurological disorder, psychological diseases; or with severe hepatic, renal or respiratory dysfunction;
5. Known or suspected liver dysfunction, including NASH, HBV or HCV-related hepatitis;
6. History of gastroscope within 1 year;

(6) Current antidepressant, steroids or NSAID use; (7) Patients who had only reflux-related symptoms or who had predominantly reflux-related symptoms; (8) Not willing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From March 2018 to August 2018 ，patient went to the Gastroenterology clinics of the second affiliated hospital of xi'an jiaotong university, Xijing Hospital, Tangdu Hospital, Xi'an No.3 Hospital, and received gastroscopy.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of organic dyspepsia. | 3 months
  To collect the results of gastroscopy in patients who meet inclusion criteria, and to calculate the incidence of organic dyspepsia to analyze the predictive value of alarm symptoms.

SECONDARY OUTCOMES:
The incidence of gastric cancer | 3 months
  To collect the results of gastroscopy in patients who meet inclusion criteria, and to calculate the incidence of gastric cancer to analyze the predictive value of alarm symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jinhai Wang, MD, Study Director — The Second Affiliated Hospital of Xi'an Jiaotong University,Xi'an, Shaanxi, China
Locations (1):
- The second affiliated hospital of xi'an jiaotong university, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei Z, Yang Q, Yang Q, Yang J, Tantai X, Xing X, Xiao C, Pan Y, Liu N, Wang J. Rome III, Rome IV, and Potential Asia Symptom Criteria for Functional Dyspepsia Do Not Reliably Distinguish Functional From Organic Disease. Clin Transl Gastroenterol. 2020 Dec;11(12):e00278. doi: 10.14309/ctg.0000000000000278. PMID 33512804
- [Derived] Wei ZC, Yang Q, Yang Q, Yang J, Tantai XX, Xing X, Xiao CL, Pan YL, Wang JH, Liu N. Predictive value of alarm symptoms in patients with Rome IV dyspepsia: A cross-sectional study. World J Gastroenterol. 2020 Aug 14;26(30):4523-4536. doi: 10.3748/wjg.v26.i30.4523. PMID 32874062